CLINICAL TRIAL: NCT02457364
Title: Prospective Observational Trial of Initial Non-operative Management of Ventral Hernia Repair
Brief Title: Non-Op Management of Ventral Hernia Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mike K Liang, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0372
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Hernia, Ventral
Keywords: non-operative management
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ventral hernias are among the most common surgical diseases among patients.The natural history of patients with ventral hernias who are managed non-operatively is unknown. The aim of this prospective trial is to document the natural history of patients who are undergoing initially non-operative management. The investigators hypothesize that 1) the risk of emergency ventral hernia repair is low, 2) the risk of elective ventral hernia repair is high, and 3) patients managed non-operatively will develop increasing hernia size and symptom progression. This is a prospective observational study of all patients undergoing non-operative management at LBJ General Hospital. Patients will be consented and then followed for 5 years. Phone interviews will be done with these patients yearly to assess surgical and medical history, information about their hernia, including pain level due to the hernia, as well as function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing initial non-operative management as chosen by current practice patterns
* All patients who opt for non-operative management due to personal choice, lack of symptoms or concerns regarding surgical risks.
* Age 18 or older

Exclusion Criteria:

* Patient meets surgery criteria but elects for surgery within 1 year due to personal scheduling
* Patient smokes < 1 pack per day, is actively quitting smoking, and desires to follow-up within 3 months upon smoking cessation
* Patient with BMI < 35 kg/m2, is actively losing weight, and desires to follow-up within 3 months upon weight loss goals being met
* Patient is unlikely to be able to follow-up due to no personal or home phone
* Patient is enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a ventral hernia who are undergoing non-operative management of their hernia at LBJ General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical repair of the ventral hernias per patient year | Once a year for 5 years

SECONDARY OUTCOMES:
Rate of emergency repair of ventral hernias per patient year | Once a year for 5 years
Rate of elective repair of ventral hernias per patient year | Once a year for 5 years
Rate of emergency room visits per patient year | Once a year for 5 years

OTHER OUTCOMES:
Change in pain from baseline using the Visual Analog Scale for Pain | Once a year for 5 years
Change in patient function from baseline using the HerQLes Survey | Once a year for 5 years
Change in patient quality of life from baseline using the HerQLes Survey | Once a year for 5 years
Change in hernia size based on clinical exam or CT scan | Once a year for 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- LBJ General Hospital-UT Health, Houston, Texas, United States

REFERENCES:
- [Background] Bedewi MA, El-Sharkawy MS, Al Boukai AA, Al-Nakshabandi N. Prevalence of adult paraumbilical hernia. Assessment by high-resolution sonography: a hospital-based study. Hernia. 2012 Feb;16(1):59-62. doi: 10.1007/s10029-011-0863-4. Epub 2011 Jul 28. PMID 21796449
- [Background] Meier DE, OlaOlorun DA, Omodele RA, Nkor SK, Tarpley JL. Incidence of umbilical hernia in African children: redefinition of "normal" and reevaluation of indications for repair. World J Surg. 2001 May;25(5):645-8. doi: 10.1007/s002680020072. PMID 11369993
- [Background] Lauscher JC, Martus P, Stroux A, Neudecker J, Behrens U, Hammerich R, Buhr HJ, Ritz JP. Development of a clinical trial to determine whether watchful waiting is an acceptable alternative to surgical repair for patients with oligosymptomatic incisional hernia: study protocol for a randomized controlled trial. Trials. 2012 Feb 7;13:14. doi: 10.1186/1745-6215-13-14. PMID 22314130
- [Background] Ah-Kee EY, Kallachil T, O'Dwyer PJ. Patient awareness and symptoms from an incisional hernia. Int Surg. 2014 May-Jun;99(3):241-6. doi: 10.9738/INTSURG-D-14-00039.1. PMID 24833146
- [Background] Bellows CF, Robinson C, Fitzgibbons RJ, Webber LS, Berger DH. Watchful waiting for ventral hernias: a longitudinal study. Am Surg. 2014 Mar;80(3):245-52. PMID 24666865
- [Background] Mudge M, Hughes LE. Incisional hernia: a 10 year prospective study of incidence and attitudes. Br J Surg. 1985 Jan;72(1):70-1. doi: 10.1002/bjs.1800720127. PMID 3155634
- [Background] Cevese PG, D'Amico DF, Biasiato R, Frego MG, Tropea A, Giaconi MA, Bianchera GG. Peristomal hernia following end-colostomy: a conservative approach. Ital J Surg Sci. 1984;14(3):207-9. PMID 6500908
- [Background] Cherney DZ, Siccion Z, Chu M, Bargman JM. Natural history and outcome of incarcerated abdominal hernias in peritoneal dialysis patients. Adv Perit Dial. 2004;20:86-9. PMID 15384802
- [Background] Eid GM, Wikiel KJ, Entabi F, Saleem M. Ventral hernias in morbidly obese patients: a suggested algorithm for operative repair. Obes Surg. 2013 May;23(5):703-9. doi: 10.1007/s11695-013-0883-5. PMID 23494458
- [Background] Liu NW, Hackney JT, Gellhaus PT, Monn MF, Masterson TA, Bihrle R, Gardner TA, House MG, Koch MO. Incidence and risk factors of parastomal hernia in patients undergoing radical cystectomy and ileal conduit diversion. J Urol. 2014 May;191(5):1313-8. doi: 10.1016/j.juro.2013.11.104. Epub 2013 Dec 10. PMID 24333109
- [Background] Marsman HA, Heisterkamp J, Halm JA, Tilanus HW, Metselaar HJ, Kazemier G. Management in patients with liver cirrhosis and an umbilical hernia. Surgery. 2007 Sep;142(3):372-5. doi: 10.1016/j.surg.2007.05.006. PMID 17723889
- [Background] Fitzgibbons RJ Jr, Ramanan B, Arya S, Turner SA, Li X, Gibbs JO, Reda DJ; Investigators of the Original Trial. Long-term results of a randomized controlled trial of a nonoperative strategy (watchful waiting) for men with minimally symptomatic inguinal hernias. Ann Surg. 2013 Sep;258(3):508-15. doi: 10.1097/SLA.0b013e3182a19725. PMID 24022443